CLINICAL TRIAL: NCT04872153
Title: Feasibility of Technology-based Cognitive-motor Training in Rehabilitation: A Pilot-trial
Brief Title: Exergames in In-patient Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eling DeBruin (Other)
Responsible Party: Sponsor-Investigator, Eling DeBruin, Prof. Dr., Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BASEC Nr. 2020-02388
Record Dates: First submitted 2021-03-29; First posted 2021-05-04 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Rehabilitation; Cardiovascular Diseases; Geriatric Patients; Parkinson Disease
Keywords: exergame; motor-cognitive training; feasibility; rehabilitation
MeSH Terms: conditions — Cardiovascular Diseases; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The patients allocated to the intervention group will conduct simultaneously combined cognitive-motor training in form of exergames using the Dividat Senso in addition to the standard rehabilitation treatment plan. Both the Dividat Senso and the training games are specifically developed considering the needs and requirements of older adults but also clinicians/therapists.
  Interventions: Behavioral: Dividat Senso Exergames
- Control Group (No Intervention): The patients of the control group follow the standard rehabilitation treatment plan including: 3x 30min physiotherapy, 8x 30min group therapy, 3x 45min group therapy (group therapy includes body- focused therapy, mindfulness therapy, respiratory therapy, gymnastics, hiking etc.)

INTERVENTIONS:
Behavioral: Dividat Senso Exergames — The intervention period in the rehabilitation setting will be equal to the length of the stay in the rehabilitation clinic (between 2-3 weeks, according to each cantonal/regional regulations and insurance coverage) and will include short daily training sessions using the Senso (5x/week à 10- 15min), resulting in 15 to 20 training sessions in total.
  Each session contains various combinations of the Dividat exergames (each of the games lasts around 2-3min).
  Arms: Intervention Group

SUMMARY:
This pilot trial aims to evaluate the feasibility and effectiveness of a technology-based intervention for cognitive-motor training in rehabilitation clinics with geriatric, neurological and cardiac patients.

The primary objective of this pilot study is to evaluate the feasibility of exergame-based cognitive-motor training in in-patient rehabilitation settings.

The secondary objective of this pilot trial is to evaluate the effectiveness of an expanded rehabilitation treatment (combining exergame training with conventional care) on physical and cognitive functioning in different patient groups.

DETAILED DESCRIPTION:
This study is a pilot trial with two arms: an intervention group where the conventional treatment during the stay in the in-patient rehabilitation clinic is extended with a technology-based cognitive-motor intervention and a control group following just the conventional treatment. Participants will be randomly allocated to one of the two groups. The selected methods to evaluate the primary and secondary endpoints include quantitative and qualitative measures. This national study will be conducted in Switzerland in a multicentre setup; three rehabilitation clinics are involved as study centres.

The study will include at least 40 patients in each of the rehabilitation clinics involved as study centres (20 patients in the intervention group, 20 patients in the control group), resulting in a total sample size of 120 patients. At clinic entry, patients potentially fulfilling all inclusion criteria will be informed in oral and written about the study and asked if they wish to participate. All interested participants will then be screened for eligibility. The included participants will then undergo a baseline assessment battery and will be subsequently randomly allocated to the intervention or the control group using a block randomization.

Screening as well as baseline measurements (T1-measurements) are conducted within the first two days upon entry at the rehabilitation clinic. T1-measurements will last around 60-70 minutes. One day after T1- measurements, the intervention will begin (for patients in the intervention group). The intervention period will be equal to the length of the stay in the rehabilitation clinic (between 2-3 weeks, according to each cantonal/regional regulations and insurance coverage) and will include short daily training sessions using the Dividat Senso (5x/week à 10-15min), resulting in 10 to 15 training sessions in total. The training sessions will be supervised by a qualified study investigator (carefully observing patients while training and also preventing/aiding in case of adverse events). At the last two days before discharge from the clinic, post-measurements (T2-measurements) will be performed with all (intervention & control) study participants. T2-measurements last around 70-80 minutes.

Intervention group:

The patients allocated to the intervention group will conduct simultaneously combined cognitive- motor training on a technological device providing exergames, the Dividat Senso. Both, the hardware (Dividat Senso) and the software (exergames) are specifically developed considering the needs and requirements of older adults but also clinicians/therapists.

The Dividat Senso is a platform for the dynamic recording of steps, weight shifts and other body movements producing forces. The platform includes 20 sensors (strain gauges), 5 vibration motors and an light-emitting diode (LED) control. It is certified as a medical device class 1 and used by clinics, hospitals and nursing and care homes in 15 countries worldwide. It is connected to a small computer (running the software) and a large screen.

The Dividat exergames specifically target all cognitive functions relevant for the successful mastering of activities of daily living such as executive and attentional functions and physical functions such as balance and coordination. The games are played by conducting body movements, mainly steps in four directions (front, right, left, back) but also body weight shifting.

The Dividat software is a web-based environment that includes data backing (Dividata), an administrative interface (Dividat Manager) and an intelligent, adaptable training environment with the exergames for motor-cognitive training (Dividat Play). In the Dividat Manager, participants can be registered as users and their training program can be managed. The training software (Dividat Play) contains an algorithm for automatic, real-time adaptation of the difficulty of a training game to the skills of a user. Moreover, the training applied in this study is progressive in the course of the intervention period; patients start with the easier games in the first week, progressing to more difficult games in the second week and so on. Therapists and study investigators have the opportunity to individually adapt the training plan to meet each patient's functional capacity in the Dividat Manager. Thus, personalized training and optimal challenge for each patient are ensured.

The intervention period in the rehabilitation setting will be equal to the length of the stay in the rehabilitation clinic (between 2-3 weeks, according to each cantonal/regional regulations and insurance coverage) and will include short daily training sessions using the Senso (5x/week à 10- 15min), resulting in 10 to 15 training sessions in total.

Each session contains various combinations of the Dividat exergames (each of the games lasts around 2-3min).

Control group:

The patients of the control group follow the standard rehabilitation procedure including per week: 3x 30min physiotherapy, 8x 30min group therapy, 3x 45min group therapy (group therapy includes body- focused therapy, mindfulness therapy, respiratory therapy, gymnastics, hiking etc.).

ELIGIBILITY:
Inclusion Criteria:

* Patients with prescription for rehabilitation*
* ≥ 50 years old
* Able to score ≥ 20 at the Mini Mental State Examination (MMSE)
* Able to provide a signed informed consent
* Physically able to stand for at least 3min without external support (self-report)

Exclusion Criteria:

* Mobility or cognitive limitations or comorbidities which impair the ability to use the training games and overall system
* Conservatively treated osteoporotic fractures
* Previous or current major psychiatric illness (e.g. schizophrenia, bipolar disorder, recurrent major depression episodes)
* History of drugs or alcohol abuse
* Terminal illness
* Severe sensory impairments (mainly visual, auditory, color blindness)
* Insufficient knowledge of German to understand the instructions/games

  * *In the rehabilitation clinics involved as study centres, mainly persons suffering from cardiovascular diseases (clinic Seewis), persons suffering from neurological diseases (esp. Parkinson's Disease according to the United Kingdom Brain Bank criteria) (clinic Zihlschlacht) and geriatric patients (clinic Dussnang) will be included in this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Adverse events are assessed during the data collection period, an average of 3 to 4 weeks.
  Related and un-related adverse events during the pre-post assessments as well as during each training session will be registered
Attrition rate | The attrition rate is assessed during the data collection period, an average of 3-4 weeks.
  Number of participants lost during the trial will be recorded (drop-outs in both groups)
Adherence rate | The adherence rate is assessed for all training sessions during the intervention period, an average of 3-4 weeks.
  Percentage of the number of attended training sessions in relation to the number of planned training sessions
System Usability Scale (SUS) | The SUS is completed at the post-measurement by the intervention group. The survey lasts 2 minutes.
  Participants of the intervention group will receive a survey form at the end of the intervention period regarding usability of the device used for the delivery of the exergame training (Dividat Senso)
Nasa Task Load Index (NASA-TLX) | The NASA-TLX is assessed after each training sessions during the intervention period. The survey lasts 1-2 minutes.
  The NASA-TLX is a self-report, multidimensional assessment tool that rates perceived workload in order to assess a task, a system, or other aspects of performance (in this case the DIVIDAT exergames). It contains five subscales: Mental Demand, Physical Demand, Temporal Demand, Performance, Effort and Frustration. A score from 1-100 is calculated based by averaging all answers to all questions.
User Experience | The questionnaire is completed at the post-measurement by the intervention group. The survey lasts 2 minutes.
  A questionnaire with (self-developed) questions regarding perceived enjoyment during training, perceived positive effects, intention to use after study's end etc. will be filled out by the intervention group
Training motivation | The question is assessed before each training session during the intervention period, an average of 3-4 weeks..
  Average training motivation based on motivation question in each session (Scale 1-5) answered by patients.

SECONDARY OUTCOMES:
Changes in psychomotor speed | Assessment takes place at pre- and post-measurement within the two days after entry respectively before discharge. The 6-RTT lasts 5 minutes.
  The Reaction Time Test (6-RTT) conducted on the Dividat Senso measures psychomotor speed in terms of reaction to visual stimuli using the lower extremities in 6 directions (front right, front left, right, left, back right & back left).
Changes in mental flexibility | Assessment takes place at pre- and post-measurement within the two days after entry respectively before discharge. The TMT lasts ca. 10 minutes.
  To assess mental flexibility (a part of executive functions), the Trail Making Test (TMT) is used pre- and post-intervention. This paper-pencil-test is resulting in a time value in seconds. Less time needed to conducted the test is related to better performance.
Changes in inhibitory control | Assessment takes place at pre- and post-measurement within the two days after entry respectively before discharge. The test lasts 10 minutes.
  To assess interference control (a part of executive functions), the Color-Word Interference Test is used pre- and post-intervention. The result is a time value measured in seconds, furthermore, errors are counted. Less time and less errors is related to better performance.
Changes in selective attention | Assessment takes place at pre- and post-measurement within the two days after entry respectively before discharge. The Go/No-Go lasts 5 minutes.
  The Go/No-Go Test conducted on the Dividat Senso measures selective attention. Participants fixate on a small grey dot in the middle of the screen. Crosses (+) and Xs (x) appear on the right and left side of the grey dot in randomised order. The task is to ignore the + and just conduct a step as quickly as possible as soon as in the direction that an x appears.
Changes in functional mobility | Assessment takes place at pre- and post-measurement within the two days after entry respectively before discharge. The TUG lasts 2 minutes.
  The Timed Up and Go (TUG) test is conducted. At the start signal participants must stand up from a chair, walk three meters at a comfortable walking speed, come back and sit down on the chair again. Time to complete the task in seconds is recorded. The use of walking aids is noted.
Changes in physical performance | Assessment takes place at pre- and post-measurement within the two days after entry respectively before discharge. The SPPB lasts 5 minutes.
  To assess physical performance the Short Physical Performance Battery (SPPB) is used resulting in a total score of 12 points with a minimum score of 0 and a maximum score of 4 for each sub-test. The SPPB consist of 3 sub-tests including a balance test (e.g. tandem stance, semi-tandem stance, single leg stance), 4-meter gait test, and 5-chair rises test. A higher score means a better balance performance.
Changes in Single-Task Walking | Assessment takes place at pre- and post-measurement within the two days after entry respectively before discharge. The Single-Task Walk lasts 3 minutes.
  Participants have to walk a 10m distance at their preferred speed and their maximal speed while still feeling safe.
Changes in Dual-Task Walking | Assessment takes place at pre- and post-measurement within the two days after entry respectively before discharge. The Dual-Task Walk lasts 3 minutes.
  Participants have to walk a 10m distance at their perferred speed while calculating serial sevens backwards.

CONTACTS AND LOCATIONS:
Overall Officials: Eling De Bruin, Prof. Dr., Principal Investigator — ETH Zurich - Institute of Human Movement Sciences and Sport
Locations (2):
- Switzerland (2):
  - Rehaklinik Dussnang, Dussnang, Thurgau
  - Rehaklinik Zihlschlacht, Zihlschlacht-Sitterdorf, Thurgau

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Jaggi S, Wachter A, Adcock M, de Bruin ED, Moller JC, Marks D, Schweinfurther R, Giannouli E. Feasibility and effects of cognitive-motor exergames on fall risk factors in typical and atypical Parkinson's inpatients: a randomized controlled pilot study. Eur J Med Res. 2023 Jan 16;28(1):30. doi: 10.1186/s40001-022-00963-x. PMID 36647177
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886